CLINICAL TRIAL: NCT05739292
Title: A Single Center, Randomized, Observer-blinded, Active Comparator Phase I Study to Assess the Safety and Immunogenicity of Meningococcal (Groups A, C, W-135, X and Y) Conjugate Vaccine in Healthy Adults Aged 19 to 55 Years Old
Brief Title: Safety and Immunogenicity of Pentavalent Meningococcal Conjugate Vaccine (EuNmCV-5) in Healthy Adults Aged 19 to 55 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EuVCT_MCV102
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-05

CONDITIONS: Infection, Meningococcal
MeSH Terms: conditions — Meningococcal Infections | interventions — Vaccines, Conjugate; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EuNmCV-5 (Experimental): Healthy adults received 0.5mL single intramuscular dose on Day 0.
  Interventions: Biological: EuNmCV-5
- Menveo (Active Comparator): Healthy adults received 0.5mL single intramuscular dose on Day 0.
  Interventions: Biological: Menveo

INTERVENTIONS:
Biological: EuNmCV-5 — 0.5mL single intramuscular dose on Day 0
  Other Names: Meningococcal(Groups A, C, W-135, X, and Y) Conjugate Vaccine
  Arms: EuNmCV-5
Biological: Menveo — 0.5mL single intramuscular dose on Day 0
  Other Names: Meningococcal(Groups A, C, Y, and W-135) Conjugate Vaccine
  Arms: Menveo

SUMMARY:
Phase I study to evaluate safety and immunogenicity in healthy adult subjects following a single dose administration of Meningococcal (Group A, C, W-135, X, and Y)-CRM197 Conjugate vaccine

ELIGIBILITY:
Inclusion Criteria:

* Subjects 19 to 55 years of age
* Written informed consent
* Available for all visits and telephone calls scheduled for the study

Exclusion Criteria:

* Previous or suspected disease caused by N. meningitides
* Household and/or intimate exposure to an individual with culture-proven N. meningitides infection within 60 days prior to screening
* Serious acute, chronic or progressive disease as determined by investigator
* History of alcohol or substance abuse

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited adverse events | within 7 days post vaccination
  local and systemic AEs
Occurrence of unsolicited adverse events | within 28 days post vaccination
Occurrence of serious adverse events | within 180 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: YJ Choi, Study Director — EuBiologics Co.,Ltd
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim Y, Bae S, Yu KS, Lee S, Lee C, Kim J, Her H, Oh J. A randomized study to evaluate the safety and immunogenicity of a pentavalent meningococcal vaccine. NPJ Vaccines. 2024 Aug 7;9(1):140. doi: 10.1038/s41541-024-00935-8. PMID 39112515